CLINICAL TRIAL: NCT06329856
Title: Exploring Indications and Practices of Administering Artificial Hydration to Terminal Cancer Patients and Establishing Clinical Consensus Guideline in Taiwan
Brief Title: Exploring Indications and Practices of Administering Artificial Hydration to Terminal Cancer Patients in Taiwan
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202301218RIND
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-03

CONDITIONS: Terminal Cancer; Hospice; Palliative Medicine
Keywords: Artificial hydration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- members of the Taiwan Academy of Hospice Palliative Medicine: members of the Taiwan Academy of Hospice Palliative Medicine
  Interventions: Behavioral: Administering of artificial hydration
- members of the Taiwan Society of Cancer Palliative Medicine: members of the Taiwan Society of Cancer Palliative Medicine
  Interventions: Behavioral: Administering of artificial hydration

INTERVENTIONS:
Behavioral: Administering of artificial hydration — Administering of artificial hydration to terminal cancer patients

SUMMARY:
Background: The issue of artificial hydration for terminal cancer patients is a classic ethical dilemma in palliative care. It is a common practice especially when patients are incapable of oral intake; however, there is a lack of research on indications and practices for the provision of artificial hydration to terminal cancer patients in Taiwan. The investigators aim to conduct a nationwide survey of palliative care physicians on their indications (general or specific), and practices of providing artificial hydration to terminal cancer patients. With that understanding of reasoning and clinical practice, the investigators would further establish an indigenous, evidence-based consensus guideline to serve as a reference for physicians in Taiwan.

Methods: The study is comprised of two parts. The first part is to conduct a nationwide survey of palliative and oncology care specialists with a questionnaire designed from literature reviews and principles of clinical ethics. After validation of the questionnaire, the investigators will e-mail it to members of the Taiwan Academy of Hospice Palliative Medicine and the Taiwan Society of Cancer Palliative Medicine. The primary outcome measure of the study is the indication and clinical practice of artificial hydration, and the secondary outcome is factors associated with the administration or withdrawal of hydration.

The second part is to establish a national consensus on clinical guidelines for administering artificial hydration, where the investigators will conduct a modified Delphi method for 6 rounds. Literature reviews will be first performed and 14 sessions of one-to-one interviews in Round 1 to develop a draft. Subsequent rounds comprise questionnaire surveys among all panelists, teleconferences and e-mail discussions among core members, and cancer patients/patients' family discussions. Statistical criteria include median and disagreement scores according to the Inter-Percentile Range Adjusted for Symmetry. Items voted for by 70% or more panelists will be selected and formalized into a consensus guideline.

Expected results: The investigators hypothesize that the indication to administer artificial hydration to the terminal cancer patient is multi-factorial and culturally based.

Conclusion: The establishment of a consensus guideline will help clinicians to make an appropriate decision from ethical, medical, cultural, and emotional factors and facilitate cancer patients to achieve a good quality of dying.

DETAILED DESCRIPTION:
Background: The issue of artificial hydration for terminal cancer patients is a classic ethical dilemma in palliative care. It is a very common practice especially when the terminal cancer patient is incapable of oral intake; however, there is a lack of research on indications and practices for the provision of artificial hydration to terminal cancer patients in Taiwan. The investigators aim to conduct a nationwide survey of palliative care physicians on their indications (general or specific), and practices of providing artificial hydration to terminal cancer patients. With that understanding of reasoning and clinical practice, the investigators would further establish an indigenous, evidence-based consensus guideline to serve as a reference for physicians in Taiwan.

Methods: The study is comprised of two parts. The first part is to conduct a nationwide survey of palliative and oncology care specialists exploring the indication and practices of administrating artificial hydration to terminal cancer patients. The questionnaire is mainly designed from literature reviews and principles of clinical ethics. After validation of the questionnaire, the investigators will e-mail it to members of the Taiwan Academy of Hospice Palliative Medicine and the Taiwan Society of Cancer Palliative Medicine. A 200 NTD equivalent voucher/gift will be provided to each respondent as an incentive. The investigators will send two follow-up e-mail reminders after two weeks apart. The primary outcome measure of the study is the indication and clinical practice of artificial hydration, and the secondary outcome is factors associated with the administration or withdrawal of hydration.

To reach an 80% response rate, 1270 out of 1589 effective members need to reply to the questionnaire. Basic demographic data will be summarized as total numbers and percentages for categorical variables. Differences in categorical variables will be compared using t-test and Chi-square tests. Cronbach's alpha values of scales are calculated to determine the internal consistency of the scales used. Logistic regressions will be applied to determine factors affecting the administration or withdrawal of artificial hydration.

The second part is to establish a national consensus on clinical guidelines for administering artificial hydration. Taking the questionnaire result as a first-hand reference, the investigators will conduct a modified Delphi method for 6 rounds to reach a final consensus. The investigators will perform literature reviews and 14 sessions of one-to-one interviews in Round 1 to develop a draft. Subsequent rounds (Round 2-6) comprise questionnaire surveys among all panelists, teleconferences and e-mail discussions among core members, and cancer patients/patients' family discussions. Statistical criteria include median score, and disagreement score according to the Inter-Percentile Range Adjusted for Symmetry. Items with a total of 70% or more panelists voting will be selected and formalized into a consensus guideline.

Expected results: The investigators hypothesize that the indication to administer artificial hydration to the terminal cancer patient is multi-factorial and culturally based.

Conclusion: The establishment of the consensus guideline will help clinicians to make the appropriate decision from ethical, medical, cultural, and emotional factors and facilitate the cancer patient to achieve a good quality of dying.

ELIGIBILITY:
Inclusion Criteria:

* Taiwan Academy of Hospice Palliative Medicine
* Taiwan Society of Cancer Palliative Medicine
* At least a year in training to take care of terminally ill patients
* Have signed informed consent.

Exclusion Criteria:

* No clinical experience in palliative care
* Decline to sign informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: From the name list of the Taiwan Academy of Hospice Palliative Medicine and Taiwan Society of Cancer Palliative Medicine
Sampling Method: Non-Probability Sample
Enrollment: 1270 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Likert scale on alteration of administer artificial hydration to the terminal cancer patient and principles of clinical ethics | Within 1 month
  Multi-factorial and culturally based questionnaire in a nationwide survey of palliative and oncology care specialist, to explore the 5- to 9-point scale of opinion on indication and practices of administrating artificial hydration to terminal cancer patients
Distributive statistics | At most 6 months
  Statistical analyses of quality indicators from 14 sessions of one-to-one interviews and questionnaire surveys among panelists, to be formalized into a consensus guideline when over 70% of panelists voting for a questionnaire item
Disagreement score according to the Interpercentile Range Adjusted for Symmetry (IPRAS) for survey results | Within 6 months
  Higher scores indicating a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yi Cheng, Study Chair — Department of Family Medicine, College of Medicine and Hospital, National Taiwan University
Locations (1):
- Department of Family Medicine, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Anonymous survey and collated data would not reflect individual personal participant data

REFERENCES:
- [Background] Chang YK, Kaplan H, Geng Y, Mo L, Philip J, Collins A, Allen LA, McClung JA, Denvir MA, Hui D. Referral Criteria to Palliative Care for Patients With Heart Failure: A Systematic Review. Circ Heart Fail. 2020 Sep;13(9):e006881. doi: 10.1161/CIRCHEARTFAILURE.120.006881. Epub 2020 Sep 9. PMID 32900233
- [Background] De Meyer D, Kottner J, Beele H, Schmitt J, Lange T, Van Hecke A, Verhaeghe S, Beeckman D. Delphi procedure in core outcome set development: rating scale and consensus criteria determined outcome selection. J Clin Epidemiol. 2019 Jul;111:23-31. doi: 10.1016/j.jclinepi.2019.03.011. Epub 2019 Mar 25. PMID 30922885
- [Result] Cheng SY, Lin CP, Chan HY, Martina D, Mori M, Kim SH, Ng R. Advance care planning in Asian culture. Jpn J Clin Oncol. 2020 Sep 5;50(9):976-989. doi: 10.1093/jjco/hyaa131. PMID 32761078
- [Result] Finkelstein EA, Bhadelia A, Goh C, Baid D, Singh R, Bhatnagar S, Connor SR. Cross Country Comparison of Expert Assessments of the Quality of Death and Dying 2021. J Pain Symptom Manage. 2022 Apr;63(4):e419-e429. doi: 10.1016/j.jpainsymman.2021.12.015. Epub 2021 Dec 22. PMID 34952169
- [Result] Welk TA. Clinical and ethical considerations of fluid and electrolyte management in the terminally ill client. J Intraven Nurs. 1999 Jan-Feb;22(1):43-7. PMID 10335177
- [Result] Schmidlin E. Artificial hydration: the role of the nurse in addressing patient and family needs. Int J Palliat Nurs. 2008 Oct;14(10):485-9. doi: 10.12968/ijpn.2008.14.10.31492. PMID 18978694
- [Result] Torres-Vigil I, Cohen MZ, de la Rosa A, Cardenas-Turanzas M, Burbach BE, Tarleton KW, Shen WM, Bruera E. Food or medicine: ethnic variations in perceptions of advanced cancer patients and their caregivers regarding artificial hydration during the last weeks of life. BMJ Support Palliat Care. 2012 Sep;2(3):276-9. doi: 10.1136/bmjspcare-2012-000205. Epub 2012 Jul 23. PMID 24654201
- [Result] Morita T, Tei Y, Inoue S. Agitated terminal delirium and association with partial opioid substitution and hydration. J Palliat Med. 2003 Aug;6(4):557-63. doi: 10.1089/109662103768253669. PMID 14516497
- [Result] Morita T, Shima Y, Miyashita M, Kimura R, Adachi I; Japan Palliative Oncology Study Group. Physician- and nurse-reported effects of intravenous hydration therapy on symptoms of terminally ill patients with cancer. J Palliat Med. 2004 Oct;7(5):683-93. doi: 10.1089/jpm.2004.7.683. PMID 15588360
- [Result] Morita T, Hyodo I, Yoshimi T, Ikenaga M, Tamura Y, Yoshizawa A, Shimada A, Akechi T, Miyashita M, Adachi I; Japan Palliative Oncology Study Group. Association between hydration volume and symptoms in terminally ill cancer patients with abdominal malignancies. Ann Oncol. 2005 Apr;16(4):640-7. doi: 10.1093/annonc/mdi121. Epub 2005 Jan 31. PMID 15684225
- [Result] Morita T, Hyodo I, Yoshimi T, Ikenaga M, Tamura Y, Yoshizawa A, Shimada A, Akechi T, Miyashita M, Adachi I; Japan Palliative Oncology Study Group. Artificial hydration therapy, laboratory findings, and fluid balance in terminally ill patients with abdominal malignancies. J Pain Symptom Manage. 2006 Feb;31(2):130-9. doi: 10.1016/j.jpainsymman.2005.06.015. PMID 16488346
- [Result] Bear AJ, Bukowy EA, Patel JJ. Artificial Hydration at the End of Life. Nutr Clin Pract. 2017 Oct;32(5):628-632. doi: 10.1177/0884533617724741. Epub 2017 Aug 16. PMID 28813202
- [Result] Bruera E, Belzile M, Watanabe S, Fainsinger RL. Volume of hydration in terminal cancer patients. Support Care Cancer. 1996 Mar;4(2):147-50. doi: 10.1007/BF01845764. PMID 8673352
- [Result] Sato K, Miyashita M, Morita T, Tsuneto S, Shima Y. End-of-Life Medical Treatments in the Last Two Weeks of Life in Palliative Care Units in Japan, 2005-2006: A Nationwide Retrospective Cohort Survey. J Palliat Med. 2016 Nov;19(11):1188-1196. doi: 10.1089/jpm.2016.0108. Epub 2016 Jul 27. PMID 27463530
- [Result] Bruera E, Hui D, Dalal S, Torres-Vigil I, Trumble J, Roosth J, Krauter S, Strickland C, Unger K, Palmer JL, Allo J, Frisbee-Hume S, Tarleton K. Parenteral hydration in patients with advanced cancer: a multicenter, double-blind, placebo-controlled randomized trial. J Clin Oncol. 2013 Jan 1;31(1):111-8. doi: 10.1200/JCO.2012.44.6518. Epub 2012 Nov 19. PMID 23169523
- [Result] Nakajima N, Takahashi Y, Ishitani K. The volume of hydration in terminally ill cancer patients with hydration-related symptoms: a prospective study. J Palliat Med. 2014 Sep;17(9):1037-41. doi: 10.1089/jpm.2013.0557. Epub 2014 Jul 22. PMID 25050699
- [Result] Wu CY, Chen PJ, Ho TL, Lin WY, Cheng SY. To hydrate or not to hydrate? The effect of hydration on survival, symptoms and quality of dying among terminally ill cancer patients. BMC Palliat Care. 2021 Jan 12;20(1):13. doi: 10.1186/s12904-021-00710-9. PMID 33435925
- [Result] Wu CY, Chen PJ, Cheng SY, Suh SY, Huang HL, Lin WY, Hiratsuka Y, Kim SH, Yamaguchi T, Morita T, Tsuneto S, Mori M; EASED Investigators. Association between the amount of artificial hydration and quality of dying among terminally ill patients with cancer: The East Asian Collaborative Cross-Cultural Study to Elucidate the Dying Process. Cancer. 2022 Apr 15;128(8):1699-1708. doi: 10.1002/cncr.34108. Epub 2022 Feb 1. PMID 35103989
- [Result] Morita T, Bito S, Koyama H, Uchitomi Y, Adachi I. Development of a national clinical guideline for artificial hydration therapy for terminally ill patients with cancer. J Palliat Med. 2007 Jun;10(3):770-80. doi: 10.1089/jpm.2006.0254. PMID 17592989
- [Result] A.S.P.E.N. Ethics Position Paper Task Force; Barrocas A, Geppert C, Durfee SM, Maillet JO, Monturo C, Mueller C, Stratton K, Valentine C; A.S.P.E.N. Board of Directors; American Society for Parenteral and Enteral Nutrition. A.S.P.E.N. ethics position paper. Nutr Clin Pract. 2010 Dec;25(6):672-9. doi: 10.1177/0884533610385429. Epub 2010 Nov 4. No abstract available. PMID 21051546
- [Result] Chiu TY, Hu WY, Cheng SY, Chen CY. Ethical dilemmas in palliative care: a study in Taiwan. J Med Ethics. 2000 Oct;26(5):353-7. doi: 10.1136/jme.26.5.353. PMID 11055038
- [Result] Chiu TY, Hu WY, Huang HL, Yao CA, Chen CY. Prevailing ethical dilemmas in terminal care for patients with cancer in Taiwan. J Clin Oncol. 2009 Aug 20;27(24):3964-8. doi: 10.1200/JCO.2008.21.4643. Epub 2009 May 26. PMID 19470919
- [Result] Huang HL, Yao CA, Hu WY, Cheng SY, Hwang SJ, Chen CD, Lin WY, Lin YC, Chiu TY. Prevailing Ethical Dilemmas Encountered by Physicians in Terminal Cancer Care Changed After the Enactment of the Natural Death Act: 15 Years' Follow-up Survey. J Pain Symptom Manage. 2018 Mar;55(3):843-850. doi: 10.1016/j.jpainsymman.2017.11.033. Epub 2017 Dec 6. PMID 29221846
- [Result] Cheng SY, Dy S, Hu WY, Chen CY, Chiu TY. Factors affecting the improvement of quality of dying of terminally ill patients with cancer through palliative care: a ten-year experience. J Palliat Med. 2012 Aug;15(8):854-62. doi: 10.1089/jpm.2012.0033. Epub 2012 Jun 27. PMID 22738375
- [Result] Lin CP, Peng JK, Chen PJ, Huang HL, Hsu SH, Cheng SY. Preferences on the Timing of Initiating Advance Care Planning and Withdrawing Life-Sustaining Treatment between Terminally-Ill Cancer Patients and Their Main Family Caregivers: A Prospective Study. Int J Environ Res Public Health. 2020 Oct 29;17(21):7954. doi: 10.3390/ijerph17217954. PMID 33138212
- [Result] Ganzini L. Artificial nutrition and hydration at the end of life: ethics and evidence. Palliat Support Care. 2006 Jun;4(2):135-43. doi: 10.1017/s1478951506060196. PMID 16903584